CLINICAL TRIAL: NCT06160427
Title: Connective Tissue Matrix (CTM) for Rotator Cuff Tendinopathy: A Randomized Controlled Trial
Brief Title: Connective Tissue Matrix for Rotator Cuff Tendinopathy
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Collaborators: Connective Tissue Matrix Biomedical, LLC (Unknown)
Responsible Party: Principal Investigator, Patrick DeMeo, MD, Professor and Institute Chair of the Department of Orthopaedic Surgery, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-264-FN
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-04

CONDITIONS: Tendinopathy; Shoulder Pain; Rotator Cuff Tendinitis; Rotator Cuff Tendinosis
Keywords: rotator cuff tendinopathy
MeSH Terms: conditions — Tendinopathy; Shoulder Pain; Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: Two-arm, double-blinded, randomized controlled trial with the primary objective of evaluating non-inferiority of CTM (study intervention arm) to PRP (active comparator arm) for rotator cuff tendinopathy pain and function.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will be randomized to one of the two arms by unblinded research personnel. Unblinded key study personnel will prepare the injection of either CTM Boost or PRP using an opaque sleeve to obscure the contents of the injection. Both patients and investigators will be blinded to treatment arm.
  Each participant will undergo an antecubital blood draw of 60 milliliers (mL). Staff will wait about 20 minutes after the blood draw to injection time. This will be done to maintain blinding due to the 17 minutes it takes for the system to produce PRP. For patients in the CTM arm, the PRP blood draw serves as a placebo draw and the specimen will be discarded afterwards, in order to maintain blinding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CTM Treatment (Experimental): 2.0 cc (cubic centimeter) dose injection of CTM Boost will be administered by injection directly into the rotator cuff using a 20 gauge needle.
  Interventions: Biological: CTM Boost
- PRP Treatment (Active Comparator): Each participant randomized to this arm will receive a single injection of Platelet Rich Plasma (PRP).
  Interventions: Biological: PRP

INTERVENTIONS:
Biological: CTM Boost — Connective Tissue Matrix (CTM) Boost is a decellularized Human Cellular and Tissue Based Allograft derived from placental connective tissue. It is considered a minimally-manipulated biologic by the FDA and is marketed as an allograft for repairing connective tissue. It is administered via injection.
  Arms: CTM Treatment
Biological: PRP — PRP is derived by a sample of blood drawn from a patient and concentrated to include mainly platelets and potent inflammatory mediators which promote healing.
  At baseline, a blood draw of 60 milliliter (mL) will be obtained and concentrated in an Angel System to yield 5 cc of PRP and a supra-physiological concentration of white blood cells. All injections will be done under ultrasound guidance. A two-part injection process will be used. An advancing 20 gauge 1.5-inch needle first placed 3 mL of 1% xylocaine proximal to the tendinopathic area or tear. The needle will then be re-inserted at the proximal aspect of the lesion and slowly removed while infiltrating of 5 mL of PRP without activation with Calcium Chloride/thrombin at the lesion and surrounding tendon.
  Arms: PRP Treatment

SUMMARY:
The purpose of this research study is to determine if the effectiveness of a single injection of CTM Boost in the treatment of patients with rotator cuff tendinopathy (RCT) is as effective as a single injection of platelet rich plasma (PRP) in reducing the symptoms of RCT.

DETAILED DESCRIPTION:
Rotator cuff tendinopathy (RCT), is a chronic degenerative process which causes both shoulder pain as well as limited range of motion. It is currently estimated that approximately 5% of RCT is being managed surgically, which highlights the importance of effective non-operative treatment strategies.

The advent of platelet rich plasma (PRP), a sample of blood drawn from a patient and concentrated to include mainly platelets and potent inflammatory mediators which promote healing, has shown promise as another treatment modality when injected at the site of tendon damage. Placenta-derived decellularized connective tissue matrix (CTM) may represent an alternative therapy for RCT. Placenta-derived biologics can be administered as an injection and have been shown to promote tenocyte proliferation and to reduce inflammation in vitro, thus potentially accelerating and enhancing tendon healing.

This study is being conducted to determine if injection of CTM Boost is non-inferior to injection of PRP with regard to pain and function at Month 6 post-injection in patients with rotator cuff tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years old with rotator cuff tendinopathy
* A PRP or CTM-type injection was determined by the clinician to be the proper medical treatment course and patient is willing to undergo the injection

Exclusion Criteria:

* Patients with adhesive capsulitis
* Patients with acromio-clavicular joint impingement, retracted tears, significant labral lesions or significant glenohumeral arthrosis
* Patients with joint instability
* History of shoulder surgery or corticosteroid injection in the past 3 months
* Patients with any medical conditions that affect healing, such as end-stage renal disease or uncontrolled diabetes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
determine if injection of CTM Boost is non-inferior to injection of PRP | 6 months
  Mean Western Ontario Rotator Cuff Index (WORC) Score The WORC has 21 items in four domains, including physical symptoms (10 questions), sports/recreation/work (4 questions), lifestyle (4 questions) and emotions (3 questions). Raw scores range from 0 to 2100, with a higher score indicating decreased quality of life because of pathological condition of the rotator cuff.

SECONDARY OUTCOMES:
Mean Western Ontario Rotator Cuff Index (WORC) Score | at 6 months
  Mean Western Ontario Rotator Cuff Index (WORC) Score The WORC has 21 items in four domains, including physical symptoms (10 questions), sports/recreation/work (4 questions), lifestyle (4 questions) and emotions (3 questions). Raw scores range from 0 to 2100, with a higher score indicating decreased quality of life because of pathological condition of the rotator cuff.
assessment of superiority of CTM to PRP (if non-inferiority established)/ WORC Score | Each visit up to 24 months
  Mean Western Ontario Rotator Cuff Index (WORC) Score The WORC has 21 items in four domains, including physical symptoms (10 questions), sports/recreation/work (4 questions), lifestyle (4 questions) and emotions (3 questions). Raw scores range from 0 to 2100, with a higher score indicating decreased quality of life because of pathological condition of the rotator cuff.
assessment of superiority of CTM to PRP (if non-inferiority established) / VAS Pain Scale | Each visit up to 24 months
  Visual Analog Scale (VAS) pain scale The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
assessment of superiority of CTM to PRP (if non-inferiority established) / SANE | Each visit up to 24 months
  Single Assessment Numeric Evaluation (SANE) The Single Assessment Numeric Evaluation (SANE) is a patient rating from 0-100. Patients rate their current illness score in relation to their pre-injury baseline. SANE scores are most commonly used by orthopedic sports specialist surgeons, and usually for the shoulder and the knee.
assessment of superiority of CTM to PRP (if non-inferiority established) / ASES | Each visit up to 24 months
  American Shoulder and Elbow Surgeons Shoulder (ASES) Score The ASES score is a 10-item measure of shoulder pain and function. Pain is assessed on a 10-cm visual analog scale (VAS) and accounts for 50% of the total score. The remaining 50% of the score is determined by the responses to 10 4-point Likert-scale questions related to physical function
assessment of superiority of CTM to PRP (if non-inferiority established) / empty can exercise | Each visit up to 24 months
  empty can exercise with dumbbell resistance (number of seconds to fatigue)
assessment of superiority of CTM to PRP (if non-inferiority established) / side laying external rotation with dumbbell resistance | Each visit up to 24 months
  Side-lying external rotation with dumbbell resistance (number of repetitions in 30 seconds)
assessment of superiority of CTM to PRP (if non-inferiority established) / full can with dumbbell resistance | Each visit up to 24 months
  Full can exercise with dumbbell resistance (number of repetitions in 60 seconds)
assessment of superiority of CTM to PRP (if non-inferiority established) / external rotation at 0 and 90 degrees | Each visit up to 24 months
  External rotation at 0 and 90 degrees with Thera-Band resistance (number of seconds to fatigue)
safety of injection of CTM boost compared to PRP | 6 months
  number of adverse events
severity of tendinopathy | 6 months
  Magnetic Resonance Imaging (MRI)-based grading scale MRIs will be scored on rubric from 0-5: 0, no tendinopathy; 1, mild tendinopathy; 2, moderate tendinopathy; 3, moderate tendinopathy + partial thickness tear present; 4, severe tendinopathy +partial thickness tear present; 5, severe tendinopathy + full thickness tear present
assessment of superiority of CTM to PRP (if non-inferiority established) | 6 months
  serum levels of inflammatory cytokines IL-1β and TNF-α as well as serum level of Fibroblast growth factor (FGF)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Demeo, MD, Principal Investigator — Allegheny Health Network
Locations (4):
- United States (4):
  - Allegheny Health Network Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Allegheny Health Network Federal North Medical Office Building, Pittsburgh, Pennsylvania
  - AHN Wexford Health & Wellness Pavilion, Wexford, Pennsylvania
  - AHN Wexford Hospital, Wexford, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] A Hamid MS, Sazlina SG. Platelet-rich plasma for rotator cuff tendinopathy: A systematic review and meta-analysis. PLoS One. 2021 May 10;16(5):e0251111. doi: 10.1371/journal.pone.0251111. eCollection 2021. PMID 33970936
- [Background] Lin MT, Wei KC, Wu CH. Effectiveness of Platelet-Rich Plasma Injection in Rotator Cuff Tendinopathy: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Diagnostics (Basel). 2020 Mar 28;10(4):189. doi: 10.3390/diagnostics10040189. PMID 32231127
- [Background] Gotoh M, Hamada K, Yamakawa H, Yanagisawa K, Nakamura M, Yamazaki H, Ueyama Y, Tamaoki N, Inoue A, Fukuda H. Interleukin-1-induced subacromial synovitis and shoulder pain in rotator cuff diseases. Rheumatology (Oxford). 2001 Sep;40(9):995-1001. doi: 10.1093/rheumatology/40.9.995. PMID 11561109
- [Background] Gotoh M, Hamada K, Yamakawa H, Nakamura M, Yamazaki H, Ueyama Y, Tamaoki N, Inoue A, Fukuda H. Perforation of rotator cuff increases interleukin 1beta production in the synovium of glenohumeral joint in rotator cuff diseases. J Rheumatol. 2000 Dec;27(12):2886-92. PMID 11128681
- [Background] Yanagisawa K, Hamada K, Gotoh M, TokunagaT, Oshika Y, Tomisawa M, Lee YH, Handa A, Kijima H, Yamazaki H, Nakamura M, Ueyama Y, Tamaoki N, Fukuda H. Vascular endothelial growth factor (VEGF) expression in the subacromial bursa is increased in patients with impingement syndrome. J Orthop Res. 2001 May;19(3):448-55. doi: 10.1016/S0736-0266(00)90021-4. PMID 11398859
- [Background] Sachinis NP, Yiannakopoulos CK, Chalidis B, Kitridis D, Givissis P. Biomolecules Related to Rotator Cuff Pain: A Scoping Review. Biomolecules. 2022 Jul 22;12(8):1016. doi: 10.3390/biom12081016. PMID 35892325
- [Background] Dean BJ, Snelling SJ, Dakin SG, Murphy RJ, Javaid MK, Carr AJ. Differences in glutamate receptors and inflammatory cell numbers are associated with the resolution of pain in human rotator cuff tendinopathy. Arthritis Res Ther. 2015 Jul 10;17(1):176. doi: 10.1186/s13075-015-0691-5. PMID 26160609
- [Background] Chen J, Svensson J, Sundberg CJ, Ahmed AS, Ackermann PW. FGF gene expression in injured tendons as a prognostic biomarker of 1-year patient outcome after Achilles tendon repair. J Exp Orthop. 2021 Mar 11;8(1):20. doi: 10.1186/s40634-021-00335-0. PMID 33694106
- [Background] Scarpone M, Rabago D, Snell E, Demeo P, Ruppert K, Pritchard P, Arbogast G, Wilson JJ, Balzano JF. Effectiveness of Platelet-rich Plasma Injection for Rotator Cuff Tendinopathy: A Prospective Open-label Study. Glob Adv Health Med. 2013 Mar;2(2):26-31. doi: 10.7453/gahmj.2012.054. PMID 24416661
- [Background] Braun C, Handoll HH. Estimating the Minimal Important Difference for the Western Ontario Rotator Cuff Index (WORC) in adults with shoulder pain associated with partial-thickness rotator cuff tears. Musculoskelet Sci Pract. 2018 Jun;35:30-33. doi: 10.1016/j.msksp.2018.02.003. Epub 2018 Feb 12. PMID 29471221
- [Background] Bushnell BD, Bishai SK, Krupp RJ, McMillan S, Schofield BA, Trenhaile SW, McIntyre LF. Treatment of Partial-Thickness Rotator Cuff Tears With a Resorbable Bioinductive Bovine Collagen Implant: 1-Year Results From a Prospective Multicenter Registry. Orthop J Sports Med. 2021 Aug 13;9(8):23259671211027850. doi: 10.1177/23259671211027850. eCollection 2021 Aug. PMID 34409115
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- See also: Sealed Envelope | Power calculator for continuous outcome non-inferiority trial — https://www.sealedenvelope.com/power/continuous-noninferior/
- See also: Daines R. LibGuides: Statistics Resources: Partial Eta Squared — https://resources.nu.edu/statsresources/eta